CLINICAL TRIAL: NCT06273189
Title: Does Ultrasonic Bone Scalpel Improve Surgical Outcomes in SSRO?
Brief Title: Ultrasonic Bone Scalpel in BSSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Selin Celebi, Resident, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/558
Record Dates: First submitted 2024-01-18; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Maxillofacial Abnormalities
Keywords: Sagittal split osteotomy; ultrasonic bone scalpel; neurosensory disturbance
MeSH Terms: conditions — Maxillofacial Abnormalities

STUDY DESIGN:
Intervention Model Description: double blind
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lindeman (Experimental): BSSO were performed with Lindeman and round bur
  Interventions: Device: Conventional
- Bone scalpel (Active Comparator): BSSO were performed unilaterally using an ultrasonic bone scalpel
  Interventions: Device: Bone Scalpel

INTERVENTIONS:
Device: Conventional — In conventional group, contralateral side mandibular osteotomies were performed with Lindeman and round bur (Karl Storz, Tuttlingen, Germany)
  Other Names: Group I
  Arms: Lindeman
Device: Bone Scalpel — In ultrasonic device group, osteotomies one side of the mandible were performed unilaterally using an ultrasonic bone scalpel (BoneScalpel; Misonix, Farmingdale, NY) with a serrated standard blade
  Other Names: Group II
  Arms: Bone scalpel

SUMMARY:
The conventional saw compared with the piezo surgery in BSSO to evaluate cutting time, surgery duration, amount of bleeding. The purpose of this study was to answers following clinical questions: Is ultrasonic bonescalpel effective osteotomy like conventional bur in BSSO? and 2) Does it reduce operative parameter like bleeding, duration, lingual split pattern? 3) Does it reduce postoperative morbidity after BSSO.

DETAILED DESCRIPTION:
The purpose of this study was to answers following clinical questions:

1) Is ultrasonic bonescalpel effective osteotomy like conventional bur in BSSO? 2) Does it reduce operative parameter like bleeding, duration, lingual split pattern? 3) Does it reduce postoperative morbidity after BSSO. Hypotheses of this study that ultrasonic bone scalpel can improve BSSO and its postoperative results due to strong cutting efficiency and soft tissue protective effect.

Surgical procedure; After removing the full thickness mucoperiosteal flap lingula was localized. In ultrasonic device group, osteotomies one side of the mandible were performed unilaterally using an ultrasonic bone scalpel (BoneScalpel; Misonix, Farmingdale, NY) with a serrated standard blade. In conventional group, contralateral side mandibular osteotomies were performed with Lindeman and round bur. Groups are selected randomly.

c- Follow up

The predictor variable was the type of instrument used for bone osteotomy. The instruments were ultrasonic bone scalpel and Lindeman bur. The main outcome variable are the cutting time and NSD. All patients were followed for 6 months.The authors used the 3dMD imaging system (3dMD, Atlanta, GA) and 3dMD Vultus software to evaluate the amount of postoperative edema.

ELIGIBILITY:
Inclusion Criteria:

* Patients are included with older than 18 years old,
* normal hemoglobin level, international normalized ratio in the average range,
* American Society of Anesthesiologists status of ASA I and II.

Exclusion Criteria:

* The exclusion criteria are neuropathic disease,
* recent use of nonsteroidal anti-inflammatory drugs and opioid derivatives,
* having preoperative signs of inflammation in the maxillofacial region,
* presence of excessive bleeding in the previous surgery,
* and allergy to drugs. All patients have given written informed consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Cutting Time | during procedure
  Length of cutting time was considered the time from the beginning the sagittal osteotomy to the end of making the vertical osteotomy line. The right and left side recorded separately.
neurosensory disturbance | up to six months
  Neuro sensory disturbance between the mental foramen and lower lip region on each side was evaluated subjectively after the operation day to a week. The examiner was blinded, and do not know which side of the mandible was randomly allocated to the experimental treatment.that was recorded by visual analog scale( VAS)

SECONDARY OUTCOMES:
The length of the procedure | during procedure
  this is recorded from mucogingival incision to the sagittal splitting in minutes by an unbiased researcher. The reason for determining this period is that the amount of mandibular movement and the degree of fixation difficulty vary, especially in facial asymmetric patients.
The splitting time | during procedure
  this is recorded for the right and left sides to determine the difficulty of splitting, respectively. If the time required to complete the splitting was less than 100 seconds, it was determined as 'easy,' between 100-200 seconds as 'medium'; if more than 200 seconds, it was determined as 'difficult.'
The pattern of the split | during procedure
  this is evaluated by cone-beam computed tomography that is classified into four types according to lingual split scale of Plooij et al
postoperative edema | up to six months
  The authors used the 3dMD imaging system (3dMD, Atlanta, GA) and 3dMD Vultus software to evaluate the amount of postoperative edema. Three-dimensional images were taken at maximum intercuspation when the lips were free and the eyes were open. The images were taken at 3 days, and at 6 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Emin Demirbaş, PhD,DDS, Study Director — Erciyes U; Yusuf Nuri Kaba, PhD,DDS, Principal Investigator — Erciyes U; Suheyb Bilge, PhD,DDS, Principal Investigator — Erciyes U; Selin Çelebi, PhD,DDS, Principal Investigator — Erciyes U
Locations (1):
- Selin Çelebi, Kayseri, Melikgazi, Turkey (Türkiye)

REFERENCES:
- [Background] Kim SG, Park SS. Incidence of complications and problems related to orthognathic surgery. J Oral Maxillofac Surg. 2007 Dec;65(12):2438-44. doi: 10.1016/j.joms.2007.05.030. PMID 18022466
- [Background] Yoshioka I, Tanaka T, Khanal A, Habu M, Kito S, Kodama M, Oda M, Wakasugi-Sato N, Matsumoto-Takeda S, Fukai Y, Tokitsu T, Tomikawa M, Seta Y, Tominaga K, Morimoto Y. Relationship between inferior alveolar nerve canal position at mandibular second molar in patients with prognathism and possible occurrence of neurosensory disturbance after sagittal split ramus osteotomy. J Oral Maxillofac Surg. 2010 Dec;68(12):3022-7. doi: 10.1016/j.joms.2009.09.046. Epub 2010 Aug 24. PMID 20739116
- [Background] Yamamoto R, Nakamura A, Ohno K, Michi KI. Relationship of the mandibular canal to the lateral cortex of the mandibular ramus as a factor in the development of neurosensory disturbance after bilateral sagittal split osteotomy. J Oral Maxillofac Surg. 2002 May;60(5):490-5. doi: 10.1053/joms.2002.31843. PMID 11988921
- [Background] Bruckmoser E, Bulla M, Alacamlioglu Y, Steiner I, Watzke IM. Factors influencing neurosensory disturbance after bilateral sagittal split osteotomy: retrospective analysis after 6 and 12 months. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Apr;115(4):473-82. doi: 10.1016/j.oooo.2012.08.454. Epub 2012 Nov 20. PMID 23182371
- [Background] Lanigan DT, Hey J, West RA. Hemorrhage following mandibular osteotomies: a report of 21 cases. J Oral Maxillofac Surg. 1991 Jul;49(7):713-24. doi: 10.1016/s0278-2391(10)80235-6. PMID 2056370
- [Background] Kohnke R, Kolk A, Kluwe L, Ploder O. Piezosurgery for Sagittal Split Osteotomy: Procedure Duration and Postoperative Sensory Perturbation. J Oral Maxillofac Surg. 2017 Sep;75(9):1941-1947. doi: 10.1016/j.joms.2017.05.003. Epub 2017 May 15. PMID 28595839
- [Background] Spinelli G, Lazzeri D, Conti M, Agostini T, Mannelli G. Comparison of piezosurgery and traditional saw in bimaxillary orthognathic surgery. J Craniomaxillofac Surg. 2014 Oct;42(7):1211-20. doi: 10.1016/j.jcms.2014.02.011. Epub 2014 Mar 20. PMID 24742747
- [Background] Vercellotti T. Technological characteristics and clinical indications of piezoelectric bone surgery. Minerva Stomatol. 2004 May;53(5):207-14. English, Italian. PMID 15263877
- [Background] Landes CA, Stubinger S, Ballon A, Sader R. Piezoosteotomy in orthognathic surgery versus conventional saw and chisel osteotomy. Oral Maxillofac Surg. 2008 Sep;12(3):139-47. doi: 10.1007/s10006-008-0123-7. PMID 18629552
- [Background] Beziat JL, Faghahati S, Ferreira S, Babic B, Gleizal A. [Intermaxillary fixation: technique and benefit for piezosurgical sagittal split osteotomy]. Rev Stomatol Chir Maxillofac. 2009 Nov;110(5):273-7. doi: 10.1016/j.stomax.2009.09.003. Epub 2009 Oct 20. French. PMID 19846184
- [Background] MCFALL TA, YAMANE GM, BURNETT GW. Comparison of the cutting effect on bone of an ultrasonic cutting device and rotary burs. J Oral Surg Anesth Hosp Dent Serv. 1961 May;19:200-9. No abstract available. PMID 13773910
- [Background] Sun C, Chen G, Fan T, Li W, Guo Z, Qi Q, Zeng Y, Zhong W, Chen Z. Ultrasonic bone scalpel for thoracic spinal decompression: case series and technical note. J Orthop Surg Res. 2020 Aug 8;15(1):309. doi: 10.1186/s13018-020-01838-9. PMID 32771031
- [Background] Al-Mahfoudh R, Qattan E, Ellenbogen JR, Wilby M, Barrett C, Pigott T. Applications of the ultrasonic bone cutter in spinal surgery--our preliminary experience. Br J Neurosurg. 2014 Jan;28(1):56-60. doi: 10.3109/02688697.2013.812182. Epub 2013 Jul 10. PMID 23841662
- [Background] Dammous S, Dupont Q, Gilles R. Three-dimensional computed tomographic evaluation of bilateral sagittal split osteotomy lingual fracture line and le fort I pterygomaxillary separation in orthognathic surgery using cadaver heads: ultrasonic osteotome versus conventional saw. J Oral Maxillofac Surg. 2015 Jun;73(6):1169-80. doi: 10.1016/j.joms.2014.12.017. Epub 2014 Dec 23. PMID 25795191
- [Background] Demirbas AE, Bilge S, Celebi S, Kutuk N, Alkan A. Is Ultrasonic Bone Scalpel Useful in Le Fort I Osteotomy? J Oral Maxillofac Surg. 2020 Jan;78(1):141.e1-141.e10. doi: 10.1016/j.joms.2019.09.021. Epub 2019 Sep 27. PMID 31669455
- [Background] Plooij JM, Naphausen MT, Maal TJ, Xi T, Rangel FA, Swennnen G, de Koning M, Borstlap WA, Berge SJ. 3D evaluation of the lingual fracture line after a bilateral sagittal split osteotomy of the mandible. Int J Oral Maxillofac Surg. 2009 Dec;38(12):1244-9. doi: 10.1016/j.ijom.2009.07.013. Epub 2009 Aug 26. PMID 19713076
- [Background] Hunsuck EE. A modified intraoral sagittal splitting technic for correction of mandibular prognathism. J Oral Surg. 1968 Apr;26(4):250-3. No abstract available. PMID 5237786
- [Background] Gleizal A, Bera JC, Lavandier B, Beziat JL. Piezoelectric osteotomy: a new technique for bone surgery-advantages in craniofacial surgery. Childs Nerv Syst. 2007 May;23(5):509-13. doi: 10.1007/s00381-006-0250-0. Epub 2007 Mar 14. PMID 17356890
- [Background] Kramer FJ, Ludwig HC, Materna T, Gruber R, Merten HA, Schliephake H. Piezoelectric osteotomies in craniofacial procedures: a series of 15 pediatric patients. Technical note. J Neurosurg. 2006 Jan;104(1 Suppl):68-71. doi: 10.3171/ped.2006.104.1.68. PMID 16509486
- [Background] Spinelli G, Mannelli G, Zhang YX, Lazzeri D, Spacca B, Genitori L, Raffaini M, Agostini T. Complex craniofacial advancement in paediatric patients: Piezoelectric and traditional technique evaluation. J Craniomaxillofac Surg. 2015 Oct;43(8):1422-7. doi: 10.1016/j.jcms.2015.07.012. Epub 2015 Aug 1. PMID 26302936
- [Background] Rana M, Gellrich NC, Rana M, Piffko J, Kater W. Evaluation of surgically assisted rapid maxillary expansion with piezosurgery versus oscillating saw and chisel osteotomy - a randomized prospective trial. Trials. 2013 Feb 17;14:49. doi: 10.1186/1745-6215-14-49. PMID 23414112
- [Background] Pagotto LEC, de Santana Santos T, de Vasconcellos SJA, Santos JS, Martins-Filho PRS. Piezoelectric versus conventional techniques for orthognathic surgery: Systematic review and meta-analysis. J Craniomaxillofac Surg. 2017 Oct;45(10):1607-1613. doi: 10.1016/j.jcms.2017.06.011. Epub 2017 Jul 1. PMID 28843403
- [Background] Schlee M, Steigmann M, Bratu E, Garg AK. Piezosurgery: basics and possibilities. Implant Dent. 2006 Dec;15(4):334-40. doi: 10.1097/01.id.0000247859.86693.ef. PMID 17172949